CLINICAL TRIAL: NCT00155935
Title: The Development of Human Immunologic Assays Specific to Folate Receptor Antigen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9261700718
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2007-08-13 (Estimated); Status verified 2004-01

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; immunotherapy; folate receptor; Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms

INTERVENTIONS:
Procedure: venous puncture

SUMMARY:
Ovarian cancer has the highest mortality rate of gynecologic malignancies and the overall 5-year survival rate of ovarian cancer is only 20-30%. Additionally, the incidence of ovarian cancer has increased in recent years in Taiwan. Ovarian cancer is indeed a disease that should be respected, however, there was very little research work focusing on it in Taiwan. Patients with ovarian cancer who have stage I disease (localized to ovaries) after optimal surgical staging do not need any adjuvant therapy. In contrast, patients with cancer spreading beyond the ovaries have median survival rates that decrease to less than (<) 10% for patients with bulky residual disease after surgery and treatment with platinum-based combination chemotherapy. In developing effective therapy for ovarian cancer, there should be a distinction between preventative and therapeutic approaches. Immunoprevention will be developed for women who are at an increased risk for the development of ovarian cancer. In contrast, immunotherapy would be used as an adjuvant to surgery or in combination with chemotherapy or other biologics such as chemoimmunotherapy or biochemoimmunotherapy. The folate receptor (FR) is expressed in some normal epithelial cells and is elevated in certain carcinomas. The FR has been reported to be selectively overexpressed in 90% of non-mucinous ovarian carcinomas. The specific epitopes of the folate receptor in the HLA-A2 haplotype have been identified. It appears that the folate receptor could be a target antigen for the immunotherapy of ovarian cancer.

Therefore the investigators would like to propose the development of folate receptor-specific immunologic assays. There are two aims in this project:

1. to develop and utilize assays to measure cytotoxic T-lymphocytes (CTLs) to folate receptors, and
2. to evaluate the folate receptor-specific immunologic responses between normal controls and ovarian cancer patients.

DETAILED DESCRIPTION:
Incidence of Ovarian Cancer

Ovarian cancer is the first mortality rate of gynecologic malignancies with an overall 5-year survival rate of only 20-30%. It became a more and more important disease in recent years and the incidence of ovarian cancer also increased in recent years in Taiwan. The lack of symptoms, difficulties in early diagnosis, insufficient accurate tumor markers, and lack of information about ovarian tumor biology contribute to the poor prognosis in ovarian cancer patients. The prognostic parameters for ovarian carcinomas are tumor stage, histologic subtype, degree of malignancy, and residual tumor after surgical treatment. However, these factors present an incomplete picture of the tumor biology of ovarian cancer and are frequently interrelated. Thus, the identification of new biologic factors predictive of individual disease course and prognosis would be extremely useful. From the above-mentioned data, ovarian cancer is indeed a disease that should be respected, however, there was very little research work focusing on it in Taiwan.

Treatment of ovarian cancer

Epithelial ovarian cancer (EOC) and extraovarian Müllerian carcinoma are similar pathologic entities that share a preference for peritoneal cavity involvement. The spread pattern of these tumors presents a challenge and unique opportunities for immunotherapy. Patients with EOC who have stage I disease (localized to ovaries) after optimal surgical staging, have a 5-year survival rate of 90%, with no significant change at 10 years. In contrast, patients with spreading beyond the ovaries have median survival rates that decrease to < 10% for patients with bulky residual disease after surgery and treatment with platinum-based combination chemotherapy. A randomized trial of first-line chemotherapy in patients with EOC with residual masses larger than 1 cm after initial surgery, showed a median survival period of 38 months for cisplatin/paclitaxel, significantly greater than 24 months for the cisplatin/cytoxan treatment arm. In an interim analysis of an equivalency trial, survival after carboplatin/paclitaxel was not worse than cisplatin/paclitaxel. Even though early diagnosis is an important goal of ongoing clinical research efforts, it is unclear whether advanced EOC starts as a multicentric process involving the ovaries and the peritoneal surface. It is now established that hereditary factors contribute to the development of EOC. Germline BRCA1 and BRCA2 mutations account for approximately 10% of all EOC. In a woman with a BRCA 1 or 2 mutation, lifetime risk for ovarian cancer ranges from 16%-44%. With the commercial availability of genetic testing for BRCA1 and BRCA2, more women are being identified as being at high risk for ovarian cancer. There are no clear guidelines on cancer prevention for these individuals. Although prophylactic oophorectomy is a reasonable option for women who have completed childbearing, these women are still at risk for developing peritoneal cancer. Clearly, other options for prevention are needed.

Immunotherapy for ovarian cancer

In developing effective immune-based strategies for EOC, there should be a distinction between preventative and therapeutic approaches. It is anticipated that immunoprevention (immunoprophylaxis) will be developed for women who are at an increased risk for the development of EOC. In contrast, immunotherapy would be used as an adjuvant to surgery or in combination with chemotherapy or other biologics as chemoimmunotherapy or biochemoimmunotherapy. Patients with undetectable disease after being restaged after chemotherapy could be considered for immunotherapy with the presumption that a majority does in fact have micrometastases. Development of effective immune-based concepts for prevention or treatment of EOC will require an understanding of tumor-immunology principles, mechanisms of action of the expanding array of immune modulating molecules, identification and characterization of tumor antigens, and determination of the microenvironment factors that could impact on the different immune-effector mechanisms. The clinical researcher has been provided with many immune directed agents, but progress on their integration into standard therapies has been somewhat slow.

Folate receptor

The folate receptor (FR), a 38 kDa membrane glycoprotein, is represented by a homologous family of glycoproteins, two of which (FR-a and FR-b) are attached to the cell surface by a glycosyl-phosphatidylinositol anchor; the third isoform (FR-) and its truncated version (FR-9) are constitutively secreted because of a lack of an efficient signal for glycosyl-phosphatidylinositol modification. FR-a is expressed in some normal epithelial cells and is elevated in certain carcinomas, whereas FR-b is a myeloid differentiation marker and is elevated in some nonepithelial malignancies. FR-9 is expressed in hematopoietic tissues. At present, FR is a major focus as a tumor target for multiple experimental approaches in cancer therapy. One novel approach uses bifunctional antibodies to target T cells to the FR on the surface of ovarian carcinoma cells. Selective growth inhibition of the tumor cells was obtained by this approach. The chimeric antibodies, which bind to both FR and either CD3 or CD28, produced impressive results in a xenogeneic model and in patients with advanced ovarian cancer. Similarly, a chimeric molecule consisting of a single-chain, Fv of anti-FR antibody and interleukin 2 was effective in inhibiting tumor growth in vivo. Alternatively, folic acid conjugates of single chain anti-T-cell receptor antibody could mobilize T-cell response against FR-rich tumors. Taking advantage of the nondestructive nature of FR-mediated internalization of folate-coupled macromolecules, cytotoxins such as momordin, Pseudomonas exotoxin, and maytansinoids were shown to produce selective killing of FR-rich cells. Furthermore, the toxicity of such conjugates was dependent upon receptor density on the cell surface. Folate-conjugated radiopharmaceuticals also appear to offer a means of tumor imaging/radiation therapy. Folate-coated liposomes were shown to selectively target FR-rich tumor cells, and selective killing of the malignant cells was obtained by encapsulating doxorubicin in the liposomes. By a similar strategy, it was possible to deliver antisense oligonucleotides against the epidermal growth factor receptor to FR-rich tumor cells. Furthermore, selective targeting of an adenoviral vector to FR-rich tumor cells has been achieved in the presence of an antibody to ablate the endogenous viral tropism. Finally, several studies have shown that FR, when expressed at high levels, could offer the preferred uptake route of novel classes of antifolate drugs that target glycineamide ribonucleotide formyltransferase and thymidylate synthase. A soluble form of FR has been detected in the serum and ascites of patients with ovarian cancer. The FR has been reported to be selectively overexpressed in 90% of non-mucinous ovarian carcinomas and in some other malignant tissues. The receptor has only been detected in a few other normal cell types, but not in normal ovarian surface epithelium. It seems that FR could be a potential target antigen for the immunotherapy of ovarian cancer.

Epitopes of folate receptor for human haplotype

The incidence of HLA-A2 haplotype is over 50% in the Western countries. The incidence of HLA-A2 haplotype is around 30% in Taiwan. The specific epitopes of the folate receptor in the HLA-A2 haplotype have been identified. They are E39 (FR, 191-199) EIWTHSTKV and E75 (FR, 245-253) LLSLALMLL, respectively. It seems that folate receptors could be a target antigen for the immunotherapy of ovarian cancer.

Our research team has focused on the development of a cancer vaccine and immunotherapy for several years. Our laboratory facilities have also been set up to evaluate the human immunologic assays for human papilloma virus type 16 E7 antigen by the grant supported from National Taiwan University Hospital. It is very important to set up various folate receptor-specific immunologic assays of human beings to evaluate the effect of cancer vaccine or immunotherapy for ovarian cancer in future clinical trials. So we would like to provide this proposal to address the development of folate receptor-specific immunologic assays in human beings. There are several aims in this project:

1. to develop and utilize assays to measure CTLs to folate receptors and,
2. to evaluate the folate receptor-specific immunologic responses between normal controls and ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian cancer patients

Ages: 10 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-01; Study Completion 2008-12

PRIMARY OUTCOMES:
To develop and utilize assays to measure CTLs to folate receptors

SECONDARY OUTCOMES:
To evaluate the folate receptor-specific immunologic responses between normal controls and ovarian cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Fang Cheng, MD, PhD, Principal Investigator — National Taiwan Univ. Hospital
Locations (1):
- National Taiwan Univ. Hospital, Taipei, Taiwan